CLINICAL TRIAL: NCT07146074
Title: Phase III Randomized Trial for High-risk Asymptomatic or Minimally Symptomatic Bone Metastases: Early Radiotherapy Versus Observation
Brief Title: Early Radiotherapy Versus Observation for High-risk Asymptomatic or Minimally Symptomatic Bone Metastases
Acronym: HERMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO23032GZA
Record Dates: First submitted 2025-07-30; First posted 2025-08-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Solid Neoplasms; Bone Metastases; Asymptomatic or Minimally Symptomatic; High Risk for Skeletal Events
Keywords: Bone metastases; Randomized; Radiotherapy; Symptomatic skeletal events; Preventive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: observational arm (Active Comparator): Patients in arm A will receive either systemic therapy or observation.
  Interventions: Drug: Systemic therapy (Standard of Care)/Observation
- Arm B: upfront radiotherapy arm (Experimental): Patients in arm B will receive preventive (upfront) radiotherapy in addition to either systemic therapy or observation.
  Interventions: Radiation: Preventive radiotherapy; Drug: Systemic therapy (Standard of Care)/Observation

INTERVENTIONS:
Radiation: Preventive radiotherapy — Either conventional radiotherapy (single dose of 8 Gy) or Stereotactic Ablative Body Radiation (either 1x20 Gy, 2x12 Gy, 3x10 Gy or 5x8 Gy) will be delivered depending on the participant's prognostic outcome.
  Arms: Arm B: upfront radiotherapy arm
Drug: Systemic therapy (Standard of Care)/Observation — It concerns systemic therapy if applicable according to the standard of care or only observation.

SUMMARY:
The goal of this clinical trial is to learn whether radiotherapy (i.e. treatment with ionizing radiation to destroy cancer cells) can prevent symptoms in patients with metastatic cancer, having high-risk bone metastases that currently result in no or only mild symptoms. High-risk bone metastases are bone metastases at high-risk of developing bone complications, such as fractures or myelum compression.

The main questions this study aims to answer are:

* Can preventive radiation of high-risk asymptomatic or minimally symptomatic bone metastases (and observation or medication) decrease the number of skeletal related events (i.e. bone complications due to bone metastases) in patients with metastatic cancer?
* Can preventive radiation of high-risk asymptomatic or minimally symptomatic bone metastases (and observation or medication) decrease the need for hospitalization related to such bone metastases, improve overall survival and (health-related) quality of life?
* What are the side effects of preventive radiation of high-risk asymptomatic or minimally symptomatic bone metastases?

Researchers will compare 2 treatment groups in order to answer the questions listed above: 1 group treated with medication or observation alone (group A) and 1 group treated with medication or observation and preventive radiotherapy (group B).

Participants will

* be screened to assess whether they are eligible to participate in the study.
* be randomized (i.e. drawn) into the 2 treatment groups mentioned above.
* be treated with preventive radiotherapy if they were drawn in treatment group B.
* need to attend follow-up visits (may be via teleconsultation) at 1, 3, 6, 12, 18 and 24 months after date of randomization during which safety and efficacy is monitored. During these follow-up visits, the general health condition of the participant is evaluated, the occurrence of any bone complication, the medications taken by the participant are registered, the degree of pain and location of the high-risk bone metastases are determined and possible side effects are registered. Furthermore, the participant needs to complete 2 questionnaires at each visit regarding his/her quality of life.

DETAILED DESCRIPTION:
It is estimated that two out of three patients with advanced cancer will develop metastases in the bones (i.e. bone metastases). Any type of cancer can spread to the bone, but the types of cancer in which the likelihood of spreading to the bone is greatest include prostate cancer, breast cancer, lung cancer, kidney cancer and skin cancer. The development of bone metastases is a serious complication of cancer that greatly affect quality of life. A large proportion of patients experience bone pain and associated reduced mobility. Bone metastases can also cause bone fractures. The growth of bone metastases in the vertebrae can lead to entrapment of the spinal cord. This is called spinal cord compression. The symptoms can range from mild (pain and a tingling sensation) to very severe (paralysis). In the English-language literature, these bone complications due to bone metastases are often indicated as skeletal-related events ("skeletal-related events"; SREs) or symptomatic skeletal-related events ("symptomatic skeletal-related events"; SSEs) when they also cause symptoms.

SSEs are defined as:

* symptomatic pathological fracture
* spinal cord compression leading to neurological deficit or pain
* Indication for palliative radiotherapy (for bone pain, cord compression or (impending) fracture)
* Indication for orthopedic surgery (for bone pain, cord compression or (impending) fracture)

When SSE occur that have a negative impact on the quality of life, these can be treated with systemic therapy, surgery or radiotherapy (RT). Scientific evidence is already available for radiotherapy as an effective treatment for patients with bone metastases causing symptoms. Recent data from an American trial suggest that also preventive radiotherapy of high-risk asymptomatic bone metastases may have a favorable effect. Hence, the aim of the HERMES study is to investigate if early preventive radiation of high-risk asymptomatic or minimally symptomatic bone metastases in patients with metastatic cancer can decrease the number of symptomatic skeletal events (SSEs) in a multi-centric randomized phase 3 trial.

A potential participant needs to sign an informed consent form before participating in the HERMES study. Participation in the HERMES study will comprise a screening period, during which the screening assessments must be completed, a treatment phase and a follow-up phase.

During the screening phase, eligibility of the patient to participate in the study will be assessed. Demographics data, Karnofsky performance score, information regarding medical history, prior medications and adverse events will be recorded. Moreover, the potential participant needs to complete questionnaires regarding his/her quality of life, characteristics of the high-risk metastases will be recorded based on imaging and a pain score will be determined for each lesion.

Eligible, consenting subjects will then be randomized (1:1) into one of two treatment arms: an observational arm (arm A) receiving systemic therapy / observation or an upfront RT arm (arm B) receiving upfront RT plus systemic therapy / observation.

During the treatment phase, RT should take place within 21 days after date of randomization for subjects in arm B. Participants of both study arms receive either systemic therapy or observation, according to the standard of care guidelines.

The follow-up phase consists of 6 follow-up visits which will take place at 1, 3, 6, 12, 18 and 24 months after date of randomization and during which safety and efficacy are monitored. More specifically, the Karnofsky performance score, concomitant medications and adverse events will be recorded at each visit. Moreover, the potential participant needs to complete questionnaires regarding his/her quality of life. Note that patients in arm B are strongly advised to receive additional preventive radiotherapy in case of appearance of new asymptomatic or minimally symptomatic high-risk bone metastases during follow-up. A maximum of 5 high-risk asymptomatic or minimally symptomatic bone metastases can be irradiated at once.

In case an SSE would occur, the assessments that should take place during the next follow-up visit, should be completed at that time point, preferably within one week. Afterwards, only survival data will be recorded on the planned FU visits until 24 months after the randomization date as well as possible occurrence of another SSE and hospitalizations related to the high-risk bone metastasis(es) until 24 months after the randomization date.

ELIGIBILITY:
Inclusion Criteria:

* I1: Histologically confirmed solid tumor malignancy (with polymetastastic spread (≥ 3 metastases))
* I2: High-risk bone metastasis(es) that is (are) asymptomatic or minimally symptomatic:

  *Asymptomatic or minimally symptomatic is defined as follows: O Numeric Pain Rating Scale (NRS) score ≤2 for the specific lesion(s)

  *High-risk is defined as follows (i.e. at least one of the following points must be applicable): O Bulky site of disease in bone (diameter ≥ 2 cm) O Disease involving the hip (acetabulum, femoral head, femoral neck), shoulder (acromion, glenoid, humeral head), or sacroiliac joints O Disease in long bones with cortical involvement of >1/3 in proportion to the diameter of the bone (humerus, radius, ulna, clavicle, femur, tibia, fibula, metacarpals, phalanges) O Disease in vertebrae of the junctional spine (C1-2, C7- T1, T12-L1, L5-S1) and/or disease with posterior element involvement or epidural extension (Bilsky epidural compression score 1a-3) [Bilsky et al]. The posterior elements of the spine consist of the pedicles, laminae, facets (articular processes), transverse processes, and the spinous process.
* I3: Number of Risk Factors (NRF) prognostic score 0-2
* I4: Age ≥ 18 years
* I5: Ability to provide informed consent (either by the patient or by a legally authorized representative)
* I6: A female participant is eligible to participate if she confirms not to be pregnant at screening, and one of the following conditions applies:

Is not a woman of child bearing potential or A woman of child bearing potential must confirm that she is not pregnant at screening and must agree to use a very effective method of birth control

Exclusion Criteria:

* E1: Previous RT to the target treatment site(s)
* E2: NRF prognostic score 3
* E3: Serious medical co-morbidities that preclude radiotherapy
* E4: Bone lesion complicated with a pathological fracture or impending pathologic fracture for which prophylactic stabilization is recommended, characterized by Mirels score of ≥9 [Mirels et al].
* E5: Spinal metastasis with SINS score >13 requiring upfront neurosurgical stabilization [Fourney et al].
* E6: More than 5 high-risk asymptomatic or minimally symptomatic metastatic bone locations
* E7: Patient already included in another clinical trial that would interfere with the HERMES clinical trial, as assessed by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Time to a symptomatic skeletal related event (SSE) in any bone metastasis or death due to any cause whichever occurs first | Measured from the date of randomization to the date when an SSE occurs in any bone metastasis, date of death due to any cause or last follow-up visit at 24 months after randomization whichever occurs first.
  Time to an SSE in any bone metastasis or death due to any cause whichever occurs first. An exception are SSE in bone metastases that were already treated with surgery or radiotherapy before study participation.

SECONDARY OUTCOMES:
Need for hospitalization related to the high-risk bone metastasis(es). | Measured from date of study randomization to last follow-up visit (24 months after randomization date), date of death of any cause or early end of participation in the study due to other reasons whichever occurs first.
  The number of hospitalizations related to the high-risk bone metastases will be compared between arm A (systemic therapy/observation) and arm B (systemic therapy/observation + upfront radiotherapy).
Overall survival (OS) | Measured from time of study randomization to date of death of any cause or last follow-up visit (24 months after randomization date) whichever occurs first
  Overall survival
Quality of life (QoL) measurement by EORTC QLQ-C15-PAL questionnaire (physical and emotional function, dyspnoea, pain, sleeping difficulties, appetite, nausea/vomiting, constipation, fatigue) | From screening until last follow-up visit (24 months after randomization date), date of death of any cause, early end of study participation due to other reason or unscheduled follow-up visit at 1 week after occurrence of an SSE whichever occurs first.
  Changes in the scores regarding physical and emotional function, dyspnoea, pain, sleeping difficulties, appetite, nausea/vomiting, constipation and fatigue over time compared to baseline as well as absolute scores will be compared between both treatment arms. The scale ranges from 1 up to 4 with a higher score representing a worse outcome.
Quality of life (QoL) measurement by EORTC QLQ-C15-PAL questionnaire (overall quality of life) | From screening until last follow-up visit (24 months after randomization date), date of death of any cause, early end of study participation due to other reason or unscheduled follow-up visit at 1 week after occurrence of an SSE whichever occurs first.
  Changes in the scores, representing the participant's overall quality of life, over time compared to baseline as well as absolute scores will be compared between both treatment arms. The scale ranges from 1 up to 7 with a higher score representing a better outcome.
Quality of life measurement by EuroQol Group EQ-5D-5L questionnaire (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). | From screening until last follow-up visit (24 months after randomization date), date of death of any cause, early end of study participation due to other reason or unscheduled follow-up visit at 1 week after occurrence of an SSE whichever occurs first.
  Changes in the scores, regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression, over time compared to baseline as well as absolute scores will be compared between both treatment arms.
Quality of life measurement by EuroQol Group EQ-5D-5L questionnaire (health "today"). | From screening until last follow-up visit (24 months after randomization date), date of death of any cause, early end of study participation due to other reason or unscheduled follow-up visit at 1 week after occurrence of an SSE whichever occurs first.
  Changes in the scores regarding health "today" over time compared to baseline as well as absolute scores will be compared between both treatment arms. The scale ranges from 0 up to 100 with a higher score representing a better outcome.
Acute and late toxicity | From time of ICF signing to last follow-up visit (24 months after randomization date), visit 1 week after occurrence of an SSE, date of death of any cause or early end of participation in the study due to other reason whichever occurs first.
  Adverse events in both study arms will be evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 . Only adverse events that are related to the bone metastatic disease or related to the radiotherapy (only for patients in arm B) will be reported in the context of the HERMES study.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Billiet, MD, PhD, Principal Investigator — Ziekenhuis aan de Stroom
Locations (8):
- Belgium (8):
  - ZAS Augustinus, Wilrijk, Antwerp
  - AZORG, Aalst
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout